CLINICAL TRIAL: NCT02649777
Title: Normal Values of Oxidative Stress, Taurine, and Related Markers
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 15-2091; UL1TR001082 (NIH)
Record Dates: First submitted 2016-01-04; First posted 2016-01-07 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Oxidative Stress
Keywords: oxidative stress

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The role of oxidative stress in disease pathology is increasingly recognized. At present, the development of biomarkers of this state is in its infancy and the availability of clinically validated assays is lacking. This study will better determine normal values for specific biomarkers of oxidative stress. It will also investigate normal values of taurine, a natural occurring oxidative stress protectant. A primary and specific application of this data is for the evaluation of oxidative stress, levels of the natural protectant taurine, and of associated inflammation in the context of cystathionine β-synthase (ClinicalTrials.gov study: Oxidative Stress Markers in Inherited Homocystinuria and the Impact of Taurine).

DETAILED DESCRIPTION:
This study is a one-time collection of blood and urine samples in healthy individuals. Subjects have to be fasting for 3 hours prior to the blood sampling. A maximum of 7.5 mLs of blood (1 and 1/5 teaspoon) and a urine sample will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Age: Over 8 years old and less than 50 years

Exclusion Criteria:

* Pregnancy: Females who are pregnant or lactating will be excluded from the study as the influence of pregnancy on the markers is not known nor is the impact of pregnancy on taurine known.
* Antioxidant use: Individuals taking taurine, over the counter energy drinks containing taurine or other high dose antioxidants such as Vitamin C or E, coenzyme Q, carotenes, selenium will be excluded as such intake will likely impact laboratory results.
* Inflammatory status:

  * Individuals who have a significant chronic illness or state that has a known or suspected marked inflammatory component or oxidative stress component will be excluded from the study as the illness will impact inflammatory markers.
  * Patients with an acute illness, which may impact inflammatory biomarkers, will be postponed for study entry until the acute illness is resolved. Entry into the study at a later day will be offered. The study visit will not be conducted within 3 weeks of the acute illness.
  * Smoking within the past 12 months will be excluded.

Ages: 8 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Healthy Individuals older than 8 years and less than 50 years
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2016-01; Primary Completion 2016-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Oxidative stress marker: TBARS | Time 0
  Single Draw for one-time analysis
Metabolite antioxidant: Taurine | Time 0
  Single Draw for one-time analysis

SECONDARY OUTCOMES:
Inflammation marker: Supper oxide dismutase (SOD) | Time 0
  Single Draw for one-time analysis
Inflammation marker: TGFβ | Time 0
  Single Draw for one-time analysis
Inflammation marker: myeloperoxidase | time 0
  Single Draw for one-time analysis
Metabolites: S-adenosylmethionine and S-adenosylhomocysteine | Time 0
  Single Draw for one-time analysis (same units)
Vascular function: Thromboxane B2 metabolites | Time 0
  Single Draw for one-time analysis (same units)
Oxidative stress: dityrosine | Time 0
  Single Draw for one-time analysis
Inflammation markers: IL1α, IL-1β, IL10, TNFα | Time 0
  Single Draw for one-time analysis; ELISA assay (same units)
Inflammation markers: cytokines: IL1α, IL-1β IL-1ra, IL6, IL8, IL17, MCP-1,MIP-1, MIP1α, MIPβ | Time 0
  Single Draw for one-time analysis; Luminex assay (same units)
Inflammation markers: cytokines: TNFα, IL4, IL10 and IL12 | Time 0
  Single Draw for one-time analysis; high sensitivity Luminex assay (same units)
Inflammation marker: high sensitivity CRP | Time 0
  Single Draw for one-time analysis

CONTACTS AND LOCATIONS:
Overall Officials: Johan LK Van Hove, MD, PhD, MBA, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No